CLINICAL TRIAL: NCT07114913
Title: Evaluation of Central Sensitization Parameters Based on Extra Median Symptom Distribution in Carpal Tunnel Syndrome: A Cross-sectional Study
Brief Title: Symptom Distribution and Pain Sensitization in Carpal Tunnel Syndrome
Status: Recruiting | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: 25/603
Record Dates: First submitted 2025-07-28; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Carpal Tunnel Syndrome; Central Sensitisation; Pain, Radiating
Keywords: carpal tunnel syndrome; central sensitization; central sensitization inventory; pressure pain threshold
MeSH Terms: conditions — Carpal Tunnel Syndrome; Pain | interventions — Nerve Conduction Studies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with Carpal Tunnel Syndrome
  Interventions: Diagnostic Test: Nerve ultrasound; Diagnostic Test: Nerve conduction studies; Diagnostic Test: Pressure pain threshold

INTERVENTIONS:
Diagnostic Test: Nerve ultrasound — Ultrasonographic evaluation of the median nerve at the carpal tunnel and adjacent levels
Diagnostic Test: Nerve conduction studies — Upper extremity nerve conduction studies including median-ulnar sensory and motor responses
Diagnostic Test: Pressure pain threshold — Pain pressure threshold is used to measure deep muscular tissue pain sensitivity.

SUMMARY:
This study aims to compare central sensitization parameters between carpal tunnel syndrome (CTS) patients with extra median symptom distribution and those with typical, median nerve-related symptoms. Extra median sensory spread, observed in some CTS patients beyond the anatomical boundaries of the median nerve, may reflect central sensitization mechanisms. Using the Central Sensitization Inventory and pressure pain threshold measurements, this study will assess whether extra median symptom patterns are associated with increased central sensitization.

DETAILED DESCRIPTION:
Carpal Tunnel Syndrome (CTS) is the most common entrapment neuropathy, typically presenting with numbness and tingling in the thumb, index, and middle fingers due to median nerve compression at the wrist. However, some patients report symptom spread beyond the median nerve distribution, involving ulnar regions of the hand, forearm, shoulder, or even scapular areas. This phenomenon, known as extra median symptom distribution, has been increasingly associated with central sensitization (CS).This study aims to compare central sensitization parameters between CTS patients with typical symptoms and those showing extra median spread. Pressure pain threshold (PPT) and Central Sensitization Inventory (CSI) scores will be used to evaluate sensitization levels. The initial hypothesis of this study was that patients with extra-median symptoms would exhibit lower PPT values and higher CSI scores, indicating greater central sensitivity. Findings may highlight the need to consider central mechanisms in CTS management and promote more personalized treatment approaches.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with carpal tunnel syndrome based on clinical and electrodiagnostic findings
* Being between 18 and 65 years of age
* Being literate
* Agreeing to participate in the study

Exclusion Criteria:

* Having a history of concomitant diabetes, systemic inflammatory disease, active infection, or malignancy
* Being <18 and >65 years of age
* Being illiterate
* Refusing to participate in the study
* Having a disease associated with neuropathic pain, such as polyneuropathy, radiculopathy, or multiple sclerosis
* History of injection or surgery for CTS within the last 6 months

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with CTS
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-06-21 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Pressure pain threshold | 3 months
  Pain pressure threshold (PPT) is used to measure deep muscular tissue sensitivity. Algometer is used in the measurement and low values are interpreted in favor of increased sensitivity.
Katz hand diagram | 3 months
  The Katz Hand Diagram is a self-reported symptom map used to support the diagnosis of Carpal Tunnel Syndrome (CTS). Patients are asked to mark areas on a standardized hand diagram where they experience pain, numbness, or tingling. This tool helps clinicians assess whether symptoms follow a median nerve distribution and is commonly used in both clinical and research settings due to its simplicity and diagnostic value.

SECONDARY OUTCOMES:
Central sensitization inventory (CSI) | 3 months
  Clinical instrument used in the diagnosis of central sensitization. A CSI part-A score of 40 and above is significant in the diagnosis. The score range is between 0 and 100, and as the score increases, the severity of sensitization symptoms increases.
Visual analog scale | 3 months
  The visual analog scale (VAS) is a validated subjective measure for pain, scored in the 0-10 range (0:no pain; 10: worst pain).
hand grip strength | 3 months
  Grip strength is a measure of muscle strength or the maximum force/tension produced by one's forearm muscles and is measured with a hand dynamometer.
Median nerve conduction studies-latency measurement | 3 months
  Latency values obtained in bilateral median motor and sensory nerve conduction studies.
Median nerve motor conduction studies-amplitude measurement | 3 months
  Amplitude values obtained in bilateral median motor nerve conduction studies.
Median nerve sensory conduction studies-amplitude measurement | 3 months
  Amplitude values obtained in bilateral median sensory nerve conduction studies.
Median nerve conduction studies- conduction velocity measurement | 3 months
  Conduction velocity values obtained in bilateral median motor and sensory nerve conduction studies.
Median nerve ultrasound cross-sectional area measurement | 3 months
  Median nerve cross-sectional area and echogenicity measurement
Median nerve ultrasound echogenicity measurement | 3 months
  Median nerve echogenicity measurement
Short form-12 | 3 months
  The 12-item Short Form Questionnaire (SF-12) is used for objective measurement of quality of life. The SF-12 provides two norm-based summary scores-Physical (PCS) and Mental (MCS)-each ranging from 0 to 100. Higher scores indicate better health, with 50 as the average based on U.S. norms.
Self Leeds Assessment of Neuropathic Symptoms and Sign (S-LANSS) | 3 months
  S-LANSS is a 7-question scale used to define pain of neuropathic origin. The score range is between 0-24 and a score of 12 points or more is in favor of the presence of neuropathic pain.
Boston Carpal Tunnel Questionnaire (BCTQ) | 3 months
  The Boston Carpal Tunnel Questionnaire (BCTQ) includes two subscales: the Symptom Severity Scale (SSS) and the Functional Status Scale (FSS). The SSS consists of 11 items, each scored from 1 (no symptoms) to 5 (very severe symptoms), resulting in a total score range of 11 to 55 and an average score range of 1.0 to 5.0. The FSS contains 8 items, also scored from 1 (no difficulty) to 5 (unable to perform), yielding a total score range of 8 to 40 and an average score range of 1.0 to 5.0. Higher scores on both subscales indicate greater symptom severity or functional limitation.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Ata, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- Sultan Abdülhamid Han Training and Research Hospital, Istanbul, Usküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data sharing not planned

REFERENCES:
- [Background] Aboonq MS. Pathophysiology of carpal tunnel syndrome. Neurosciences (Riyadh). 2015 Jan;20(1):4-9. PMID 25630774
- [Background] Zanette G, Cacciatori C, Tamburin S. Central sensitization in carpal tunnel syndrome with extraterritorial spread of sensory symptoms. Pain. 2010 Feb;148(2):227-236. doi: 10.1016/j.pain.2009.10.025. Epub 2009 Dec 8. PMID 20004060
- [Background] Sobeeh MG, Ghozy S, Elshazli RM, Landry M. Pain mechanisms in carpal tunnel syndrome: a systematic review and meta-analysis of quantitative sensory testing outcomes. Pain. 2022 Oct 1;163(10):e1054-e1094. doi: 10.1097/j.pain.0000000000002566. Epub 2021 Dec 15. PMID 35050958
- [Background] Woolf CJ. Central sensitization: implications for the diagnosis and treatment of pain. Pain. 2011 Mar;152(3 Suppl):S2-S15. doi: 10.1016/j.pain.2010.09.030. Epub 2010 Oct 18. PMID 20961685
- [Background] Fernandez-de-las-Penas C, de la Llave-Rincon AI, Fernandez-Carnero J, Cuadrado ML, Arendt-Nielsen L, Pareja JA. Bilateral widespread mechanical pain sensitivity in carpal tunnel syndrome: evidence of central processing in unilateral neuropathy. Brain. 2009 Jun;132(Pt 6):1472-9. doi: 10.1093/brain/awp050. Epub 2009 Mar 31. PMID 19336461
- [Background] Feng B, Gong C, You L, Lin Y, Wang Y, Ip WY, Wang Y. Central Sensitization in Patients with Chronic Pain Secondary to Carpal Tunnel Syndrome and Determinants. J Pain Res. 2023 Dec 19;16:4353-4366. doi: 10.2147/JPR.S441786. eCollection 2023. PMID 38145037